CLINICAL TRIAL: NCT04532736
Title: Comparison of Methylprednisolone or Methotrexate With Standard Treatment in the Maintenance Treatment of Medically and Surgically Treated Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Comparison of Methylprednisolone or Methotrexate in the Maintenance Treatment of Nasal Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yesim Tuncok, Pharmacologist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 216S871
Record Dates: First submitted 2019-01-15; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Nasal Polyposis
Keywords: Nasal polyposis; chronic rhinosinusitis; methotrexate; methylprednisolone; phase 2 clinical trial; mometasone furoate
MeSH Terms: conditions — Nasal Polyps | interventions — Methotrexate; Methylprednisolone; Mometasone Furoate; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: A Randomized, Controlled, Triple Armed, Parallel, Open-label Phase 2 Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methotrexate (Experimental): 10 mg Emthexate, PO, once a week during 8 weeks
  Interventions: Drug: Emthexate
- Methylprednisolone (Active Comparator): 8 mg/day Prednol, PO, for 8 weeks
  Interventions: Drug: Prednol
- Control (Active Comparator): 200 mcg/day, intranasal mometasone furoate, for 8 weeks
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Emthexate — After randomization, the patients were divided into three groups including 14 volunteers in each study groups and 11 in the control group. One of the study groups was take methotrexate (n=14, eight weeks) and the other was take methylprednisolone (n=14, eight week)
  Other Names: Methotrexate
  Arms: Methotrexate
Drug: Prednol — After randomization, the patients were divided into three groups including 14 volunteers in each study groups and 11 in the control group. One of the study groups was take methotrexate (n=14, eight weeks) and the other was take methylprednisolone (n=14, eight week)
  Other Names: Methylprednisolone
  Arms: Methylprednisolone
Drug: Mometasone Furoate — After randomization, the patients were divided into three groups including 14 volunteers in each study groups and 11 in the control group. One of the study groups was take methotrexate (n=14, eight weeks) and the other was take methylprednisolone (n=14, eight week)
  Other Names: Corticosteroid
  Arms: Control

SUMMARY:
Chronic rhinosinusitis with nasal polyposis (CRwNP) is an inflammatory disease of the nasal mucosa. It is presented with severe stuffiness, nasal discharge, facial pressure/pain, and sleep disorders. It leads to severe inconvenience to social life and the quality of life. The first step standard medical therapy consists of the topical intranasal or systemic corticosteroids. Surgery should be considered in the case of medical treatment failure. However, the recurrences are common after both surgery and medical therapies in severe disease and usually require revision surgeries or high dose corticosteroid regimens. On the contrary, either the revision surgeries or the high dose corticosteroid therapies are not capable of preventing the recurrences, treatment failures. Besides, revision surgeries usually lead to high complication rates and high dose corticosteroids usually cause severe adverse effects. The use of the short course topical intranasal corticosteroids after the surgery is generally advocated for these patients. However, the recurrence rates are still high. Hence a new and effective maintenance treatment algorithm with no severe adverse effects is required.

The hypothesis of the clinical trial is an estimated symptom recovery and superiority in both efficacy and safety by the use of low-dose methylprednisolone or methotrexate as compared to the standard maintenance therapy in treatment-resistant CRwNP patients. Therefore, the results of the present study are believed to provide data on novel maintenance therapy and suggest an alternative to the topical intranasal corticosteroids or the high-risk revision surgery.

DETAILED DESCRIPTION:
Methotrexate, as an anti-inflammatory drug used in animal experiments, and low dose systemic corticosteroid treatments have recently been suggested for the treatment of the CRwNP. Despite the several case reports of methotrexate being used for the severe and treatment-resistant CRwNP, the literature is a lack of clinical trials. Likewise, low-dose corticosteroid regimens have not been tested well contrary to the high dose corticosteroid therapy in the same course of the disease. Therefore, the main purpose of this study is to compare a low-dose of methylprednisolone or a low dose of methotrexate treatments with the standard intranasal, topical corticosteroid treatment in human volunteers with medical and surgical treatment-resistant CRwNP.

The present study was planned as a randomized, controlled, triple armed, parallel, open-label phase 2 clinical trial which is conducted in the Department of Otorhinolaryngology at Dokuz Eylül University Hospital. Human volunteers with CRwNP who are resistant to the medical and surgical therapies were recruited to the study. After randomization, the patients were divided into three groups including 14 volunteers in each study groups and 13 in the control group. One of the study groups was take methotrexate (n=14, eight weeks) and the other was take methylprednisolone (n=14, eight weeks). Each patient were evaluated by endoscopic examination, the nasal air-flow, the smell threshold, and the blood biochemistry both before and after the medications.

Efficacy goals of the study are located at below:

1. Primary efficacy variable: Lund-Kennedy endoscopic grading system (NPS)
2. Secondary efficacy variables: Total visual analog scale (VAS) score; the Turkish version of the Sinonasal Outcome Test-22 (SNOT-22); sum score of the peak nasal inspiratory flow (PNIF) and butanol olfactory threshold test (BuOT) obtained from bilateral nasal cavities; serum total immunoglobulin E (IgE) level; and the presence of peripheral eosinophilia (PE, > 500/mcl) in blood samples.

Safety goal of the study was evaluated by the examination of the adverse event reports and the number of patients who experienced adverse events.

Statistical analysis: The normality of the continuous variables was evaluated by the Shapiro Wilk test. Comparison of age was performed using one-way analysis of variance (ANOVA). Repeated measurements in three groups were analyzed using repeated measures ANOVA for 3×3 model with a within and a between-subjects factor. The results were assessed with a 95% confidence interval and at the p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of chronic rhinosinusitis with nasal polyposis (CRS) with nasal polyposis which does not respond to maintenance treatment with topical nasal corticosteroid treatment after medical and surgical treatment,
* 18-75 years of age from both sexes,
* Signed an informed consent form,

Exclusion Criteria:

* Systemic oral methylprednisolone or systemic oral methotrexate treatment for another reason,
* Has a known malignant disease,
* Have contraindications or allergies to the use of excipients in oral methotrexate or preparations,
* Contraindications or allergies in the use of oral methylprednisolone or excipients contained in the preparation,
* Have contraindications or allergies to the use of excipients contained in nasal topical mometasone furoate or its preparation,
* Pregnancy status,
* Having a pregnancy plan,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Lund-Kennedy endoscopic grading system (NPS) | Change from baseline NPS at 4th and 8th weeks visits
  Occurrence of polyps, edema, discharge, scar and crusting parameters were scored according to the 0-1-2 rating system.

SECONDARY OUTCOMES:
Total visual analog scale (VAS) | Change from baseline VAS at 4th and 8th weeks visits
  Smell, nasal discharge, nasal obstruction, facial pressure, and headache were scored between 0 (no complaint) and 10 (most annoying)
Sinonasal Outcome Test-22 (SNOT-22) | Change from baseline SNOT-22 at 4th and 8th visits
  Change in the 22-item symptom questionnaire scale used to evaluate the presence of symptoms of chronic rhinosinusitis and their effect on quality of life
Peak nasal inspiratory flow (PNIF) | Change from baseline PNIF at 4th and 8th visits
  During inspiration, nasal peak airflows were detected with the nasal mask attached to the Clement-Clark peak flow-meter. Right and left nostrils of each patient were evaluated separately.
Butanol olfactory threshold test (BuOT) | Change from baseline BuOT at 4th and 8th visits
  The odor thresholds of the patients who smelled the bottle containing 9 different concentrations of butanol between 0.00061 and 4% were determined.
Total immunoglobulin E (IgE) level | Change from baseline total IgE level at 4th and 8th visits
  To detect serum IgE level in the blood IgE level measured in peripheral blood
Presence of peripheral eosinophilia (PE, > 500/mcl) in blood samples | Change from baseline presence of peripheral eosinophilia at 4th and 8th visits
  Detection of eosinophil count> 500 / mcl in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Tuncok, MD, Principal Investigator — Dokuz Eylul University School of Medicine
Locations (1):
- Dokuz Eylul University School of Medicine, Izmir, General, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No